CLINICAL TRIAL: NCT01243268
Title: A Regulatory Requirement Post-Marketing Surveillance Study to Monitor the Safety and Efficacy of Twynsta (Telmisartan + Amlodipine SPC, q.d.) in Korean Hypertensive Patients Requiring Combination Therapy
Status: Completed | Type: Observational
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Other Study IDs: 1235.40
Record Dates: First submitted 2010-11-17; First posted 2010-11-18 (Estimated); Results first posted 2018-10-22 (Actual); Last update posted 2018-10-22 (Actual); Status verified 2017-12

CONDITIONS: Hypertension
MeSH Terms: conditions — Hypertension | interventions — telmisartan amlodipine combination

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Patients with essential hypertension
  Interventions: Drug: Twynsta tablet

INTERVENTIONS:
Drug: Twynsta tablet — Telmisartan and Amlodipine T40/A5, T80/A5 and T40/A10

SUMMARY:
This is a prospective, observational, open-label, multi-center study, which will provide detailed information about the safety and efficacy of Twynsta tablets in Korean hypertensive patients requiring combination therapy. This will present a convenient treatment option for hypertension in Korean patients.

DETAILED DESCRIPTION:
Study Design:

PMS Observational study

ELIGIBILITY:
Inclusion criteria:

No specific inclusion and exclusion criteria will be provided due to the exploratory character of the study. Patients who have initiated Twynsta tablets according to the recommended and approved usage in Korea will be consecutively enrolled.

Exclusion criteria:

No specific inclusion and exclusion criteria will be provided due to the exploratory character of the study. Patients who have initiated Twynsta tablets according to the recommended and approved usage in Korea will be consecutively enrolled.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Korean patients wtih essential hypertension
Sampling Method: Probability Sample
Enrollment: 674 (Actual)
Dates: Start 2010-12-21 (Actual); Primary Completion 2016-06-27 (Actual); Study Completion 2016-08-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Boehringer Ingelheim, Study Chair — Boehringer Ingelheim
Locations (1):
- NISND Center, One Or Multiple Sites, South Korea

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Case report forms of subjects were retrieved from 34 investigators at 26 institutions
Pre-assignment Details: The study initiated on Dec 21, 2010, but the local health authority fixed the study period as August 19, 2010 to August 18, 2016
Groups:
- Twynsta® Tablets: Subjects who received Twynsta tablets (40/5 mg, 40/10 mg, and 80/5 mg) once daily orally with water.
  Twynsta is a fixed dose combination drug composed of Telmisartan and Amlodipine.
Period: Overall Study
Arm/Group | Twynsta® Tablets
Started | 674
Completed | 610
Not Completed | 64
Not completed — Lost to Follow-up | 4
Not completed — Protocol Violation | 51
Not completed — Deviation with contract date | 7
Not completed — Duplicate subject | 2

BASELINE CHARACTERISTICS:
Population: Subjects data collected during the surveillance period (19 Aug 2010 to 18 Aug 2016).
Arm/Group | Twynsta® Tablets
Number analyzed (Participants) | 610
Age, Continuous [Mean (Standard Deviation); unit: years] | 61.96 (12.43)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 271
  Male | 339

OUTCOME MEASURES:

1. Secondary Outcome: Percentage of Subjects Who Had Achieved Normal Blood Pressure (Systolic Blood Pressure (SBP)/ Diastolic Blood Pressure (DBP) < 140/90 mmHg)
Description: Percentage of subjects who had achieved normal blood pressure (SBP/DBP < 140/90 millimeters of mercury (mmHg))is presented
Time Frame: 8±2 weeks
Population: An efficacy assessment was carried out for 531 subjects out of the 610 subjects in the safety assessment, excluding 70 subjects who had not recorded the mean sitting blood pressure (SBP, DBP) before or after the administration of the study drug and 9 subjects who had been administered the study drug for a duration shorter than 6 weeks (42 days)
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Twynsta® Tablets
Number analyzed (Participants) | 531
percentage of participants | 74.95 [71.04 to 78.58]

2. Primary Outcome: Percentage of Subjects With Adverse Events
Description: Percentage of subjects with adverse events is presented. Results are reported for short term surveillance (8±2 weeks) and Long term surveillance (16±2 weeks)
Time Frame: Short term surveillance (8±2 weeks) and Long term surveillance (16±2 weeks)
Population: Subjects data collected during the surveillance period (19 Aug 2010 to 18 Aug 2016).
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Twynsta® Tablets
Number analyzed (Participants) | 610
percentage of participants
  Short term surveillance | 3.28 [1.43 to 6.36]
  Long term surveillance | 3.80 [0.79 to 10.70]

3. Secondary Outcome: Percentage of Subjects Who Achieved DBP Response (Defined as Mean Sitting DBP < 90 mmHg or a Reduction of Over 10 mmHg)
Description: Percentage of subjects who achieved DBP response (defined as mean sitting DBP < 90 mmHg or a reduction of over 10 mmHg) is presented
Time Frame: 8±2 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Twynsta® Tablets
Number analyzed (Participants) | 531
percentage of participants | 89.45 [86.52 to 91.93]

4. Secondary Outcome: Percentage of Subjects Who Achieved SBP Response (Defined as Mean Sitting SBP < 140 mmHg or a Reduction of Over 10 mmHg)
Description: Percentage of subjects who achieved SBP response (defined as mean sitting SBP < 140 mmHg or a reduction of over 10 mmHg) is presented
Time Frame: 8±2 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Twynsta® Tablets
Number analyzed (Participants) | 531
percentage of participants | 87.76 [84.67 to 90.42]

5. Secondary Outcome: Percentage of Subjects With Diabetes or Renal Impairment Who Achieved SBP/DBP < 130/80 mmHg.
Description: Percentage of subjects with diabetes or renal impairment who achieved SBP/DBP < 130/80 mmHg is presented
Time Frame: 8±2 weeks
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: percentage of participants
Arm/Group | Twynsta® Tablets
Number analyzed (Participants) | 531
percentage of participants | 39.53 [31.04 to 48.52]

ADVERSE EVENTS:
Time Frame: Adverse events collected during the surveillance period (19 Aug 2010 to 18 Aug 2016); up to 313 weeks
Arm/Group | Twynsta® Tablets
Serious Adverse Events (participants affected / at risk) | 3/610
Other Adverse Events (participants affected / at risk) | 0/610
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Twynsta® Tablets (N=610)
Cerebral infarction (Nervous system disorders) | 1
Cardiac failure congestive (Cardiac disorders) | 1
Hepatocellular carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Boehringer Ingelheim (BI) acknowledges that investigators have the right to publish the study results. Investigators shall provide BI with a copy of any publication or presentation for review prior to any submission. Such review will be done with regard to proprietary information, information related to patentable inventions, medical, scientific, and statistical accuracy within 60 days. BI may request a delay of the publication in order to protect BI's intellectual property rights.